CLINICAL TRIAL: NCT00412360
Title: Multi-center, Open Label, Randomized Trial Comparing Single Versus Double Umbilical Cord Blood (UCB) Transplantation in Pediatric Patients With High Risk Leukemia and Myelodysplasia (BMT CTN #0501)
Brief Title: Single vs Double Umbilical Cord Blood Transplants in Children With High Risk Leukemia and Myelodysplasia (BMT CTN 0501)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0501; 2U01HL069294 (NIH); 5U24CA076518 (NIH); NCT00429598 (obsolete NCT alias)
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome; Natural Killer Cell Lymphoblastic Leukemia/Lymphoma
Keywords: Double cord blood
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma | interventions — Whole-Body Irradiation; Cyclophosphamide; fludarabine; fludarabine phosphate; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single Cord Blood Transplant (Experimental): Unrelated donor, single umbilical cord blood unit transplant; conditioning regimen: Total Body Irradiation/cyclophosphamide/fludarabine; GVHD prophylaxis: Cyclosporine A/Mycophenolate Mofetil
  Interventions: Biological: Single Umbilical Cord Blood Unit Transplant; Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Cyclosporine A; Drug: Mycophenolate Mofetil
- Double Cord Blood Transplant (Experimental): Unrelated donor, double umbilical cord blood unit transplant; Conditioning regimen: Total Body Irradiation/cyclophosphamide/fludarabine; GVHD prophylaxis: Cyclosporine A/Mycophenolate Mofetil
  Interventions: Biological: Double Umbilical Cord Blood Unit Transplant; Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Cyclosporine A; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Biological: Single Umbilical Cord Blood Unit Transplant — Unrelated donor, single umbilical cord blood unit; conditioning regimen: TBI/cyclophosphamide/fludarabine; GVHD prophylaxis: cyclosporine/MMF
  Arms: Single Cord Blood Transplant
Biological: Double Umbilical Cord Blood Unit Transplant — Unrelated donor, double umbilical cord blood unit; Conditioning regimen: TBI/cyclophosphamide/fludarabine; GVHD prophylaxis: cyclosporine/MMF
  Arms: Double Cord Blood Transplant
Radiation: Total Body Irradiation — The TBI will be delivered from either a linear accelerator or cobalt source at a dose rate of between 4 and 26 cGy/minute using energies of between 1 and 25 MV.
  Other Names: TBI
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day will be administered as a 2 hour intravenous infusion with a high volume fluid flush on Days -3 and -2.
  Other Names: Cytoxan®
Drug: Fludarabine — Fludarabine 25 mg/m2/day will be administered over 30-60 minutes intravenous infusion on Days -10 through -8. Fludarabine will not be dose adjusted for body weight.
  Other Names: Fludara
Drug: Cyclosporine A — CSA will be administered beginning on Day -3 and doses will be adjusted to maintain a level of 200-400 ng/mL by TDX method (or 100-250 ng/mL by Tandem MS or equivalent level for other CSA testing methods). CSA can be administered per institutional practice.
  Other Names: CSA
Drug: Mycophenolate Mofetil — MMF will be given at a dose of 1 gram IV q 8 hours if > 50 kg or 15 mg/kg IV q 8 hours if < 50 kg beginning the morning of Day -3.
  Other Names: MMF, Cellcept®

SUMMARY:
This study is a Phase III, randomized, open-label, multi-center, prospective study of single umbilical cord blood (UCB) transplantation versus double UCB transplantation in pediatric patients with hematologic malignancies.

DETAILED DESCRIPTION:
BACKGROUND:

In nearly every large single center or registry analysis of outcomes after UCB transplantation, cell dose is identified as an important factor influencing the incidence and rate of hematopoietic recovery, risk of transplant-related mortality, and probability of survival. Pilot data suggest that infusion of two partially human leukocyte antigen (HLA)-matched UCB units, which always augments the graft cell dose, is safe and may improve neutrophil recovery and survival. To determine whether the infusion of two UCB units enhances survival, a multi-center, open-label, randomized trial is proposed. As adequate single UCB units can be identified for more than 80% of pediatric recipients (in contrast to less than 30% for adults), this study will be open only to pediatric patients. The population will be restricted to patients with high-risk hematologic malignancy, the most common indication of UCB transplantation in children.

DESIGN NARRATIVE:

Participants will include patients 1 to 21 years of age with a diagnosis of hematological malignancy and with two partially HLA-matched UCB units. Units must be HLA-matched at 3 of 6 HLA-A and B (intermediate resolution molecular typing) and DRB1 (high resolution molecular typing) with each other and 4 of 6 with the recipient. Two appropriately HLA-matched units must be available such that one unit delivers a pre-cryopreserved, nucleated cell dose of at least 2.5 x 10^7 per kilogram and the second unit delivers at least 1.5 x 10^7 per kilogram.

Patients will be randomized no more than 14 days prior to initiation of conditioning. UCB units will be shipped prior to initiation of conditioning.

The preparative regimen will consist of the following:

* Fludarabine: 25 mg/m2/day IV on Days -10, -9, and -8.
* Total Body Irradiation (TBI): 165 cGy twice daily on Days -7, -6, -5, and -4.
* Cyclophosphamide: 60 mg/kg/day x 2 on Days -3 and -2.
* Day 0 will be the day of the UCB transplant. The Graft-vs-Host-Disease (GVHD) prophylaxis regimen will be mycophenolate mofetil (MMF) 15 mg/kg IV BID on Day -3 to Day + 45 and cyclosporine A (CSA) to maintain level 200-400 ng/mL beginning on Day -3.

Patients will be followed for at least 24 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Two partially HLA-matched UCB units. Units must be HLA-matched minimally at 4 of 6 HLA-A and B (at intermediate resolution by molecular typing) and DRB1 (at high resolution by molecular typing) loci with the patient, and the units must be HLA-matched at 3 of 6 HLA- A, B, DRB1 loci with each other (using same resolution of molecular typing as indicated above). Two appropriately HLA-matched units must be available such that one unit delivers a pre-cryopreserved nucleated cell dose of at least 2.5 x 10^7 per kilogram and the second unit at least 1.5 x 10^7 per kilogram.
* Acute myelogenous leukemia (AML) at the following stages:

  1. High risk first complete remission (CR1), defined as the following:

     * Having preceding myelodysplasia (MDS)
     * High risk cytogenetics (high risk cytogenetics: del (5q) -5, -7, abn (3q), t (6;9) complex karyotype [at least 5 abnormalities],)the presence of a high FLT3 ITD-AR (> 0.4)
     * Requiring more than 1 cycle of chemotherapy to obtain complete remission (CR);
     * FAB M6
  2. Second or greater CR
  3. First relapse with less than 25% blasts in bone marrow
  4. Morphologic complete remission with incomplete blood count recovery
* Therapy-related AML for which prior malignancy has been in remission for at least 12 months
* Acute lymphocytic leukemia (ALL) at the following stages:

  1. High risk first remission, defined as one of the following conditions:

     * Philadelphia chromosome-positive adult lymphoblastic leukemia (Ph+ ALL)
     * Mixed lineage leukemia (MLL) rearrangement with slow early response (defined as having M2 [5-25% blasts] or M3 [more than 25% blasts on bone marrow examination on Day 14 of induction therapy])
     * Hypodiploidy (less than 44 chromosomes or DNA index less than 0.81)
     * End of induction M3 bone marrow
     * End of induction M2 with M2-3 at Day 42
     * Evidence of minimal residual disease (MRD). If a patient's only high risk criterion is MRD, approval by a protocol chair or protocol officer is required for enrollment. For COG centers, this will only be for MRD greater than 1 percent by flow MRD at the end of extended induction.
  2. High risk second remission, defined as one of the following conditions:

     * Philadelphia chromosome-positive adult lymphoblastic leukemia (Ph+ ALL)
     * Bone marrow relapse less than 36 months from induction
     * T-lineage relapse at any time
     * Very early isolated central nervous system (CNS) relapse (6 months from diagnosis)
     * Slow reinduction (M2-3 at Day 28) after relapse at any time
     * Evidence of minimal residual disease (MRD). If a patient's only high risk criterion is MRD, approval by a protocol chair or protocol officer is required for enrollment. For COG centers, this will only be for MRD greater than 1 percent by flow MRD at the end of extended induction.
  3. Any third or subsequent CR
* NK cell lymphoblastic leukemia in any CR
* Biphenotypic or undifferentiated leukemia in any CR or if in first relapse must have less than 25% blasts in bone marrow (BM)
* Myelodysplastic syndrome (MDS) at any stage
* Chronic myelogenous leukemia (CML) in chronic or accelerated phase
* All patients with evidence of CNS leukemia must be treated and be in CNS CR to be eligible for study.
* Patients 16 years old or older must have a Karnofsky score of at least 70% and patients younger than 16 years old must have a Lansky score of at least 70%.
* Patients with adequate physical function as measured by:

  1. Cardiac: Left ventricular ejection fraction greater than 40% or shortening fraction greater than 26%
  2. Hepatic: Bilirubin no more than 2.5 mg/dL; alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) no more than 5 times the upper limit of normal (ULN)
  3. Renal: Serum creatinine within normal range for age, or if serum creatinine is outside normal range for age, then renal function (creatinine clearance or GFR) greater than 70 mL/min/1.73 m^2
  4. Pulmonary: Diffusing capacity of the lung for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1), or forced vital capacity (FVC) greater than 50% of predicted value (corrected for hemoglobin); if unable to perform pulmonary function tests, then O2 saturation greater than 92% of room air

Exclusion Criteria:

* Pregnant (β-positive human chorionic gonadotropin [HCG]) or breastfeeding
* Evidence of HIV infection or HIV positive serology
* Current uncontrolled bacterial, viral, or fungal infection (currently taking medication and progression of clinical symptoms)
* Autologous transplant less than 12 months prior to enrollment
* Prior autologous transplant for the disease for which the UCB transplant will be performed
* Prior allogeneic hematopoietic stem cell transplant
* Active malignancy other than the one for which the UCB transplant is being performed within 12 months of enrollment
* Inability to receive TBI
* Requirement of supplemental oxygen
* HLA-matched related donor able to donate

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 224 (Actual)
Dates: Start 2006-12; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research
Locations (38):
- United States (36):
  - University of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Childrens Hospital at Oakland, Oakland, California
  - UCSD/Rady Childrens Hospital, San Diego, California
  - University of California, San Francisco (Peds), San Francisco, California
  - The Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Nemours Childrens Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Louisville/Kosiar Children's Hospital, Louisville, Kentucky
  - Children's of New Orleans, New Orleans, Louisiana
  - DFCI/Children's Hospital of Boston, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute/Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Childrens Medical Center, Fort Worth, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Utah BMT/University of Utah Medical School, Salt Lake City, Utah
  - Virgina Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Children's Hospital at Westmead, Westmead, New South Wales, Australia
- BC Cancer Agency, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Findings were published in a manuscript.
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Shulman HM, Sullivan KM, Weiden PL, McDonald GB, Striker GE, Sale GE, Hackman R, Tsoi MS, Storb R, Thomas ED. Chronic graft-versus-host syndrome in man. A long-term clinicopathologic study of 20 Seattle patients. Am J Med. 1980 Aug;69(2):204-17. doi: 10.1016/0002-9343(80)90380-0. PMID 6996481
- [Result] Wagner JE Jr, Eapen M, Carter S, Wang Y, Schultz KR, Wall DA, Bunin N, Delaney C, Haut P, Margolis D, Peres E, Verneris MR, Walters M, Horowitz MM, Kurtzberg J; Blood and Marrow Transplant Clinical Trials Network. One-unit versus two-unit cord-blood transplantation for hematologic cancers. N Engl J Med. 2014 Oct 30;371(18):1685-94. doi: 10.1056/NEJMoa1405584. PMID 25354103
- See also: National Marrow Donor Program — https://www.nmdp.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Single UCB Transplant: Single Cord Blood Unit Transplantation: Unrelated donor, single cord blood unit
- Double UCB Transplant: Double Cord Blood Unit Transplantation: Unrelated donor, double cord blood unit
Period: Overall Study
Arm/Group | Single UCB Transplant | Double UCB Transplant
Started | 113 | 111
Completed | 112 | 108
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Not Transplanted | 1 | 2

BASELINE CHARACTERISTICS:
Population: Analysis based on intent-to-treat.
Groups:
- Single UCB Transplant: Single Umbilical Cord Blood Unit Transplantation
- Double UCB Transplant: Double Umbilical Cord Blood Unit Transplantation
- Total: Total of all reporting groups
Arm/Group | Single UCB Transplant | Double UCB Transplant | Total
Number analyzed (Participants) | 113 | 111 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (5.1) | 10.4 (5.1) | 10.4 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 41 | 96
  Male | 58 | 70 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 20 | 42
  Not Hispanic or Latino | 88 | 88 | 176
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 80 | 85 | 165
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 12 | 7 | 19
Primary Disease [Count of Participants; unit: Participants]
  Acute Myelogenous Leukemia (AML) | 39 | 38 | 77
  Acute Lymphoblastic Leukemia (ALL) | 61 | 58 | 119
  Acute Biphenotypic Leukemia | 6 | 2 | 8
  Acute Undifferentiated Leukemia | 1 | 0 | 1
  Myelodysplastic Syndrome (MDS) | 5 | 13 | 18
  Chronic Myelogenous Leukemia (CML) | 1 | 0 | 1
AML Disease Status [Count of Participants; unit: Participants] — Population: Participants with AML
  Participants
    number analyzed (Participants) | 39 | 38 | 77
    First Complete Remission (CR) | 17 | 14 | 31
    Second or Later CR | 16 | 19 | 35
    First Relapse | 1 | 3 | 4
    Morphologic CR before Complete-Blood-Count Recover | 2 | 2 | 4
    Secondary or Therapy-related | 3 | 0 | 3
ALL Disease Status [Count of Participants; unit: Participants] — Population: Participants with ALL
  Participants
    number analyzed (Participants) | 61 | 58 | 119
    First Complete Remission (CR) | 19 | 19 | 38
    Second CR | 29 | 28 | 57
    Subsequent CR | 13 | 10 | 23
    Morphologic CR before Complete-Blood-Count Recover | 0 | 1 | 1
Acute Biphenotypic Leukemia Disease Status [Count of Participants; unit: Participants] — Population: Participants with Acute Biphenotypic Leukemia
  Participants
    number analyzed (Participants) | 6 | 2 | 8
    First Complete Remission (CR) | 5 | 1 | 6
    Second CR | 1 | 1 | 2
MDS Disease Status [Count of Participants; unit: Participants] — RAEB1: Blast percentage of 5-10%; RAEB2: Blast percentage of 11-20% Population: Participants with MDS
  Participants
    number analyzed (Participants) | 5 | 13 | 18
    Refractory Anemia | 2 | 0 | 2
    Refractory Cytopenia with Multilineage Dysplasia | 2 | 3 | 5
    Refractory Anemia with Excess Blasts 1 (RAEB1) | 0 | 3 | 3
    Refractory Anemia with Excess Blasts 2 (RAEB2) | 0 | 4 | 4
    Unclassified | 1 | 3 | 4
Karnofsky Performance Score [Count of Participants; unit: Participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  Participants
    100% | 58 | 57 | 115
    90% | 38 | 43 | 81
    80% | 13 | 9 | 22
    70% | 4 | 2 | 6
Recipient CMV Status [Count of Participants; unit: Participants]
  Positive | 58 | 66 | 124
  Negative | 51 | 39 | 90
  Inconclusive | 1 | 1 | 2
  Unknown | 3 | 5 | 8
Weight at Infusion [Mean (Standard Deviation); unit: kilograms] | 39.6 (20.2) | 38.7 (19.2) | 39.15 (19.7)
Recipient to First Cord Blood Unit HLA Match [Count of Participants; unit: Participants] — Population: Transplanted participants
  Participants
    number analyzed (Participants) | 112 | 108 | 220
    3/6 | 1 | 2 | 3
    4/6 | 44 | 33 | 77
    5/6 | 51 | 59 | 110
    6/6 | 16 | 14 | 30
Recipient to Second Cord Blood Unit HLA Match [Count of Participants; unit: Participants] — Population: Double UCB transplant participants
  Participants
    number analyzed (Participants) | 0 | 108 | 108
    3/6 |  | 1 | 1
    4/6 |  | 43 | 43
    5/6 |  | 43 | 43
    6/6 |  | 21 | 21
Recipient to First Cord Blood Unit ABO Match [Count of Participants; unit: Participants] — Blood type matching between recipient and cord blood unit Population: Transplanted participants
  Participants
    number analyzed (Participants) | 112 | 108 | 220
    Major Mismatch | 30 | 25 | 55
    Minor Mismatch | 24 | 35 | 59
    Bidirectional Mismatch | 10 | 8 | 18
    No Mismatch | 44 | 36 | 80
    Unknown | 4 | 4 | 8
Recipient to Second Cord Blood Unit ABO Match [Count of Participants; unit: Participants] — Blood type matching between recipient and cord blood unit Population: Double UCB transplant participants
  Participants
    number analyzed (Participants) | 0 | 108 | 108
    Major mismatch |  | 31 | 31
    Minor mismatch |  | 29 | 29
    Bidirectional mismatch |  | 4 | 4
    No mismatch |  | 38 | 38
    Unknown |  | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Survival
Description: Overall survival is defined as survival of death from any cause.
Time Frame: 1 year post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 113 | 111
percentage of participants | 73 [63 to 80] | 65 [56 to 74]
Statistical Analysis 1: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in overall survival at one year post-randomization between participants receiving single- and double-unit cord blood transplant. The targeted sample size of 110 participants per treatment group was sufficient to maintain a type I error rate of 5% and provide more than 86% power to detect an increase in overall survival from 57% among participants receiving a single unit graft to 77% for those receiving a double-unit graft; Test type: Superiority; p = 0.17, Log Rank — Testing was performed at a significance level of 0.05

2. Secondary Outcome: Percentage of Participants With Disease-free Survival
Description: Disease-free survival is defined as survival without relapse of the primary disease.
Time Frame: 1 year post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 113 | 111
percentage of participants | 70 [60 to 77] | 64 [54 to 72]
Statistical Analysis 1: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in disease-free survival at one year post-randomization between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.11, Log Rank — Testing was performed at a significance level of 0.05

3. Secondary Outcome: Percentage of Participants With Neutrophil and Platelet Engraftment
Description: Neutrophil engraftment is defined as achieving an absolute neutrophil count greater than 500x10^6/liter for three consecutive measurements on different days. The first of the three days will be designated the day of neutrophil engraftment. Platelet engraftment is defined as achieving platelet counts greater than 50,000/microliter for consecutive measurements over 7 days without requiring platelet transfusions. The first of the 7 days will be designated the day of platelet engraftment. Subjects must not have had platelet transfusions during the preceding 7 days.
Time Frame: Days 42 and 100
Population: Transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 112 | 108
percentage of participants
  Neutrophil Engraftment at Day 42 | 89 [83 to 95] | 88 [82 to 94]
  Platelet Engraftment at Day 100 | 76 [68 to 85] | 65 [56 to 74]
Statistical Analysis 1: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in the cumulative incidence of neutrophil engraftment between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.29, Gray's test — Testing was performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in the cumulative incidence of platelet engraftment between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.04, Gray's test — Testing was performed at a significance level of 0.05

4. Secondary Outcome: Time to Neutrophil and Platelet Engraftment
Description: Platelet engraftment is defined as achieving platelet counts greater than 50,000/microliter for consecutive measurements over 7 days without requiring platelet transfusions. The first of the 7 days will be designated the day of platelet engraftment. Subjects must not have had platelet transfusions during the preceding 7 days.
Time Frame: 2 years post-transplant
Population: Transplanted participants
Measure: Median (Full Range); unit: days
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 112 | 108
days
  Neutrophil Engraftment | 21 [11 to 62] | 23 [11 to 133]
  Platelet Engraftment | 58 [28 to 295] | 84 [22 to 716]

5. Secondary Outcome: Percentage of Participants With Acute Graft-versus-host Disease (GVHD)
Description: Acute GVHD is graded according to the scoring system proposed by Przepiorka et al.1995:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area
  2. Rash on 25-50% of body surface area
  3. Rash on > 50% of body surface area
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level)*:
  0: <2 mg/dL
  1. 2-3 mg/dL
  2. 3.01-6 mg/dL
  3. 6.01-15.0 mg/dL
  4. >15 mg/dL
  GI stage*:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus * If multiple etiologies are listed for liver or GI, the organ system is downstaged by 1.
  GVHD grade:
  0: All organ stages 0 or GVHD not listed as an etiology I: Skin stage 1-2 and liver and GI stage 0 II: Skin stage 3 or liver or GI stage 1 III: Liver stage 2-3 or GI stage 2-4 IV: Skin or liver stage 4
Time Frame: Day 100 post-randomization
Population: Transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 112 | 108
percentage of participants
  Acute GVHD Grade II-IV | 57 [48 to 67] | 56 [47 to 65]
  Acute GVHD Grade III-IV | 13 [7 to 20] | 23 [15 to 31]
Statistical Analysis 1: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in the cumulative incidence of Grade II-IV acute GVHD between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.78, Gray's test — Testing was performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in the cumulative incidence of Grade III-IV acute GVHD between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.02, Gray's test — Testing was performed at a significance level of 0.05

6. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: Incidences of chronic GVHD will be graded per Shulman et al. 1980. This reference categorizes chronic GVHD as either limited or extensive. For this outcome, participants developing either type are considered to have a chronic GVHD event.
Time Frame: 1 year post-randomization
Population: Transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 112 | 108
percentage of participants
  Chronic GVHD | 30 [22 to 39] | 32 [23 to 40]
  Extensive Chronic GVHD | 9 [4 to 14] | 15 [8 to 22]
Statistical Analysis 1: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in the cumulative incidence of chronic GVHD between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.51, Gray's test — Testing was performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in the cumulative incidence of extensive chronic GVHD between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.05, Gray's test — Testing was performed at a significance level of 0.05

7. Secondary Outcome: Number of Infections Per Participant
Time Frame: 2 years post-randomization
Population: Transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 112 | 108
Participants
  0 | 10 | 9
  1 | 15 | 13
  2 | 12 | 15
  3 | 19 | 10
  4 | 17 | 15
  5 | 7 | 12
  6-10 | 19 | 24
  More than 10 | 13 | 10

8. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse is defined by either morphological or cytogenetic evidence of AML, ALL, CML, or MDS consistent with pre-transplant features. Testing for recurrent malignancy in the blood, marrow or other sites will be used to assess relapse after transplantation.
Time Frame: 1 year post-randomization
Population: Transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 112 | 108
percentage of participants | 12 [6 to 18] | 14 [7 to 21]
Statistical Analysis 1: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in the cumulative incidence of relapse between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.12, Gray's test — Testing was performed at a significance level of 0.05

9. Secondary Outcome: Percentage of Participants With Treatment-related Mortality
Description: Treatment related mortality is defined as death without relapse of the primary disease.
Time Frame: 1 year post-randomization
Population: Transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 112 | 108
percentage of participants | 19 [11 to 26] | 22 [14 to 30]
Statistical Analysis 1: Comparison: Single UCB Transplant vs Double UCB Transplant; The null hypothesis is that there is no difference in the cumulative incidence of treatment-related mortality between participants receiving single- and double-unit cord blood transplant; Test type: Superiority; p = 0.43, Gray's test — Testing was performed at a significance level of 0.05

10. Secondary Outcome: Number of Participants With Engraftment Syndrome
Time Frame: Day 100 post-transplant
Population: Transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | Single UCB Transplant | Double UCB Transplant
Number analyzed (Participants) | 112 | 108
Participants | 11 | 7

ADVERSE EVENTS:
Time Frame: 2 years post-transplant
Description: Serious Adverse Events (AE) are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected grades 3-5 adverse events were required to be reported through the AE system per protocol.
Arm/Group | Single UCB Transplant | Double UCB Transplant
Serious Adverse Events (participants affected / at risk) | 5/112 | 14/108
Other Adverse Events (participants affected / at risk) | 0/112 | 0/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single UCB Transplant (N=112) | Double UCB Transplant (N=108)
Hemolytic anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Congestive heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Respiratory failure from Pneumonia
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Acute intracranial Hemorrage (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Seizure/aspiration Pneumonia (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary Hemorrage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-03-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT00412360/Prot_SAP_ICF_000.pdf